CLINICAL TRIAL: NCT05241301
Title: Perspectives of Family Carers of Older People From Turkish and Moroccan Origin in Flanders and Brussels, Belgium, on Advance Care Planning: An Exploratory Interview Study
Brief Title: Perspectives of Family Carers of Older People From Turkish and Moroccan Origin in Belgium on Advance Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACP2021M&T
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-05

CONDITIONS: Advance Care Planning; Ethnic Minorities; Family Caregivers

STUDY DESIGN:
Intervention Model Description: one to one interviews
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One to one interviews with family carers of older people from Turkish and Moroccan origin (Other): one to one interviews
  Interventions: Other: one to one interviews

INTERVENTIONS:
Other: one to one interviews — one to one interviews to explore the perspective of family carers of older adults of Turkish and Moroccan origin in Flanders and Brussels, Belgium, concerning advance care planning (ACP)

SUMMARY:
In this study, we will explore the perspective of family carers of older adults from Turkish and Moroccan origin in Flanders and Brussels, Belgium, concerning advance care planning (ACP), more specifically concerning their knowledge about ACP, their experiences with and their points of view on ACP for their family member and their own preferences regarding how to be involved in the process of ACP for their relatives.

DETAILED DESCRIPTION:
Whether or not someone wants to engage in ACP, is often the result of a complex interplay of meanings, events, processes and assumptions constructed by the patient and is best approached by qualitative methods. Semi-structured interviews will be used in order to explore the respondents' knowledge about and experience with ACP, also their views concerning ACP for their relatives and how do they prefer to engage in the process of ACP for their relatives will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Family carers of older adults with a Turkish or a Moroccan origin who have participated in our previous studies with NCT03930823 and NCT04335214, as identified by the older adults as the most significant family carer. Older adults in our previous studies were men and women, all 65 years and older and living in Flanders and Brussels.
* and who live in Belgium and are 18 years or older and fluent in French or Dutch language.
* and who have also given informed consent to participate in this qualitative interview study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Knowledge of family carers of older adults from Turkish and Moroccan origin about advance care planning | 12 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions: Have you ever heard of advance care planning? Does that term mean anything to you? What do you know about communicating wishes in advance to family members or doctor and notice this?

SECONDARY OUTCOMES:
Experiences of family carers of older adults from Turkish and Moroccan origin have with engaging in the process of ACP for their relatives | 12 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions: Have you personally already spoken with some of your relatives about their future wishes what matters to him/her regarding his/her healthcare? If No: why? If yes: how?

OTHER OUTCOMES:
Family carers from Turkish and Moroccan origin views regarding their relatives engaging in the process of ACP? | 12 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions: Do you think it would be important that your relative discusses his/her wishes with someone? Can you explain it more in detail?
How do family carers of older adults with Turkish and Moroccan origin prefer to engage in the process of ACP for their relatives? | 12 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions: What do you think about speaking openly with your relative about ACP? Who do you think should be involved? Which role do you want in this process?
  * What do you hope this conversation will bring about? What are your expectations? What would you like to discuss? - Would you need help to start this conversation? Or would you record this alone?

CONTACTS AND LOCATIONS:
Overall Officials: Hakki Demirkapu, MD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Faculteit Geneeskunde en Farmacie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirkapu H, Edally W, De Vleminck A, Van den Block L, De Maesschalck S, Devroey D. Views on advance care planning of family members of older adults with Turkish and Moroccan backgrounds: An exploratory interview study. Palliat Med. 2024 Oct;38(9):1000-1009. doi: 10.1177/02692163241261207. Epub 2024 Jun 25. PMID 38916263